CLINICAL TRIAL: NCT03217149
Title: Heliox for Neonate With Acute Respiratory Distress Syndrome (ARDS): A Randomized Controlled Trial
Brief Title: Heliox for Neonate With Acute Respiratory Distress Syndrome (ARDS)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Daping Hospital and the Research Institute of Surgery of the Third Military Medical University (Other)
Responsible Party: Principal Investigator, Ma Juan, Principal Investigator, Daping Hospital and the Research Institute of Surgery of the Third Military Medical University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: heliox for ARDS
Record Dates: First submitted 2017-07-12; First posted 2017-07-13 (Actual); Last update posted 2017-07-13 (Actual); Status verified 2017-07

CONDITIONS: ARDS

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- heliox combined with mechanical ventilation (MV) (Experimental): heliox combined with mechanical ventilation (MV) is given to infant with ARDS
  Interventions: Drug: heliox combined with MV
- mechanical ventilation (Active Comparator): mechanical ventilation (MV) is given to infant with ARDS
  Interventions: Drug: MV

INTERVENTIONS:
Drug: heliox combined with MV — heliox combined with MV is given to infant with ARDS
  Arms: heliox combined with mechanical ventilation (MV)
Drug: MV — MV is given to infant with ARDS
  Arms: mechanical ventilation

SUMMARY:
Acute respiratory distress syndrome (ARDS) in neonates has been defined, the role of heliox is not clear.This study aimed to determine whether ARDS neonate would benefit from heliox when oxygenation deteriorated on mechanical ventilation and to identify any potential risk factors related to mortality.

DETAILED DESCRIPTION:
Acute respiratory distress syndrome (ARDS) can result in severe hypoxemia refractory to mechanical ventilation, mechanical ventilation including high frequency oscillation ventilation is the main method. But it is partial unuseful.

ELIGIBILITY:
Inclusion Criteria:

1. infant less than 28 days
2. diagnosis of ARDS
3. informed parental consent has been obtained

Exclusion Criteria:

1. major congenital malformations or complex congenital heart disease
2. transferred out of the neonatal intensive care unit without treatment

Ages: 30 Minutes to 28 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 200 (Estimated)
Dates: Start 2017-09-01 (Estimated); Primary Completion 2020-08-30 (Estimated); Study Completion 2020-08-30 (Estimated)

PRIMARY OUTCOMES:
death | within 100 days
  death

SECONDARY OUTCOMES:
Bayley Scales of Infant Development | at 2 months old and 2 years old
  the survival is assessed by Bayley Scales of Infant Development

CONTACTS AND LOCATIONS:
Overall Officials: Shi Yuan, PhD,MD, Study Director — Daping Hospital and the Research Institute of Surgery of the Third Military Medical University
Locations (1):
- Department of Pediatrics, Daping Hospital, Third Military Medical University, Chongqing, Chongqing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided